CLINICAL TRIAL: NCT02018159
Title: An Explorative Prospective Observational Study to Describe Morphokinetic De-selection Parameters in Human Embryos
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000102
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Menotropins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women treated with Menopur: Women treated with Menopur can participate with more than one cycle. 700 cycles will be enrolled.
  Interventions: Drug: menotropin

INTERVENTIONS:
Drug: menotropin
  Other Names: Menopur

SUMMARY:
This post-marketing, multi-center prospective study will be conducted in a open-label, non-interventional setting, for women seeking fertility treatment and will describe morphokinetic de-selection parameters in human embryos.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-45 years
* In Vitro Fertilisation/Intra Cytoplasmic Sperm Injection treatment in long or short protocol
* Receiving follicle stimulation with Menopur 600/1200 IU

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women seeking fertility treatment
Sampling Method: Non-Probability Sample
Enrollment: 738 (Actual)
Dates: Start 2014-01; Primary Completion 2016-02-12 (Actual); Study Completion 2016-05-12 (Actual)

PRIMARY OUTCOMES:
Incidence of direct cleavage from 1 to 3 and from 2 to 5 cells | 1 week after oocyte retrieval
Incidence of uneven blastomeres at the 2 and 4 cell stage | 1 week after oocyte retrieval
Incidence of bi- and multinucleation at 2 cell and 4 cell stage | 1 week after oocyte retrieval
Incidence of Smooth Endoplasmatic Reticulum at the Metaphase II stage, the Pro Nuclei stage and the 2, 3 and 4 cell stage | 1 week after oocyte retrieval

SECONDARY OUTCOMES:
Positive serum human Chorion Gonadotrophin (hCG) rate | 13-15 days after transfer
Implantation rate | 5 weeks after transfer
Clinical pregnancy rate | 7 weeks after transfer
Ongoing pregnancy rate | 10 weeks after transfer
Live birth rate | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Fertilitetsklinikken Hospitalsenheden Horsens, Regionshospitalet Horsens (there may be other sites in this country), Horsens, Denmark